CLINICAL TRIAL: NCT06061783
Title: Correction of Hypernatremia by Intravenous Hypotonic Solution Compared to Enteral Water, Randomized Clinical Trial
Brief Title: Correction of Hypernatremia by Intravenous Hypotonic Solution Compared to Enteral Water
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Jonathan Samuel Chavez Iñiguez, Head of nephrology Dr. Jonathan Samuel Chavez Iñiguez, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Correction of hypernatremia
Record Dates: First submitted 2023-09-20; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Hypernatremia
Keywords: Hypernatremia; intravenous hypotonic solution; enteral water
MeSH Terms: conditions — Hypernatremia | interventions — Hypotonic Solutions

STUDY DESIGN:
Intervention Model Description: Open Label randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous hypotonic solution (Active Comparator): In this group, the administration will be according to the presence of basal hyperglycemia on the day before the assignment (>180mg/dL).
  If hyperglycemia is present, it will be glucose solution 5% 500ml + injectable water 500ml intravenous every 8 hours for a total of 3,600ml daily.
  If there is no hyperglycemia, it will be 5% glucose solution 1,200ml every 8 hours for a total of 3,600ml per day.
  Interventions: Drug: Hypotonic Solution
- Enteral water (Placebo Comparator): This group will receive bottled water through the nasogastric or orogastric tube at a dose of 150 ml/hour for a total of 3,600 ml per day.
  Interventions: Drug: Water Purified

INTERVENTIONS:
Drug: Hypotonic Solution — Intravenous administration of 5% glucose solution 1,200ml every 8 hours for a total of 3,600ml per day.
  If hyperglycemia is present, it will be glucose solution 5% 500ml + injectable water 500ml intravenous every 8 hours for a total of 3,600ml daily.
  Arms: Intravenous hypotonic solution
Drug: Water Purified — administration of bottled water through the nasogastric or orogastric tube at a dose of 150 ml/hour for a total of 3,600 ml per day.
  Arms: Enteral water

SUMMARY:
Hypernatremia, defined as an elevation of serum sodium >145 mEq/L, is one of the most common electrolyte disturbances in hospitalized patients and intensive care units.

In this study, the investigator aims, for the first time, to compare two strategies used for the correction of hypernatremia, using intravenous hypotonic solution compared to naso- or orogastric tube enteral water.

DETAILED DESCRIPTION:
Hypernatremia, defined as an elevation of serum sodium >145 mEq/L, is one of the most common electrolyte disturbances in hospitalized patients and intensive care units, increasing mortality. Currently, the most effective correction strategy for hypernatremia (intravenous hypotonic solution compared to enteral water) is still a matter of debate due to a lack of evidence and clinical trials.

This study aims to determine whether the administration of intravenous hypotonic solution is more effective in the correction of hypernatremia compared to enteral water by naso- or orogastric tube. Therefore, the investigator proposes the first randomized clinical trial, which compares two strategies used for the correction of hypernatremia, with this we will determine which of the two is more effective, and we will also compare the speed of correction, renal function during hospitalization with serum creatinine and we will evaluate its safety.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with hypernatremia (serum sodium>145mEq/L).

Exclusion Criteria:

* Age below 18 years
* Pregnant, on dialysis
* Unwilling to participate or without informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The efficiency of intravenous hypotonic solution for the correction of hypernatremia compared with enteral water. | every 12 hours during the first 48hrs of treatment and then every 24 hours for the first 5 days of the study.
  Correction of hypernatremia is <145mEq/L serum sodium

SECONDARY OUTCOMES:
mortality | the first 5 days of the study
renal function | the first 5 days of the study
  serum creatinine
volume overload | the first 5 days of the study
  volume overload determined by accumulated water balance in milliliters
neurological alterations | the first 5 days of the study
  neurological disorders defined as the presence of altered state of consciousness, seizures and/or cerebral edema

OTHER OUTCOMES:
hyperglycemia, glucose >180mg/dL | the first 5 days of the study
  hyperglycemia defined as capillary glucose >180mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Samuel Chavez Iñiguez, Principal Investigator — HCG

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Polderman KH, Schreuder WO, Strack van Schijndel RJ, Thijs LG. Hypernatremia in the intensive care unit: an indicator of quality of care? Crit Care Med. 1999 Jun;27(6):1105-8. doi: 10.1097/00003246-199906000-00029. PMID 10397213
- [Background] Lindner G, Funk GC, Schwarz C, Kneidinger N, Kaider A, Schneeweiss B, Kramer L, Druml W. Hypernatremia in the critically ill is an independent risk factor for mortality. Am J Kidney Dis. 2007 Dec;50(6):952-7. doi: 10.1053/j.ajkd.2007.08.016. PMID 18037096
- [Background] Darmon M, Timsit JF, Francais A, Nguile-Makao M, Adrie C, Cohen Y, Garrouste-Orgeas M, Goldgran-Toledano D, Dumenil AS, Jamali S, Cheval C, Allaouchiche B, Souweine B, Azoulay E. Association between hypernatraemia acquired in the ICU and mortality: a cohort study. Nephrol Dial Transplant. 2010 Aug;25(8):2510-5. doi: 10.1093/ndt/gfq067. Epub 2010 Feb 17. PMID 20167570
- [Background] O'Donoghue SD, Dulhunty JM, Bandeshe HK, Senthuran S, Gowardman JR. Acquired hypernatraemia is an independent predictor of mortality in critically ill patients. Anaesthesia. 2009 May;64(5):514-20. doi: 10.1111/j.1365-2044.2008.05857.x. PMID 19413821
- [Background] Chand R, Chand R, Goldfarb DS. Hypernatremia in the intensive care unit. Curr Opin Nephrol Hypertens. 2022 Mar 1;31(2):199-204. doi: 10.1097/MNH.0000000000000773. PMID 34939612
- [Background] Thongprayoon C, Cheungpasitporn W, Petnak T, Ghamrawi R, Thirunavukkarasu S, Chewcharat A, Bathini T, Vallabhajosyula S, Kashani KB. The prognostic importance of serum sodium levels at hospital discharge and one-year mortality among hospitalized patients. Int J Clin Pract. 2020 Oct;74(10):e13581. doi: 10.1111/ijcp.13581. Epub 2020 Jun 23. PMID 32510711
- [Background] Robertson GL. Diabetes insipidus: Differential diagnosis and management. Best Pract Res Clin Endocrinol Metab. 2016 Mar;30(2):205-18. doi: 10.1016/j.beem.2016.02.007. Epub 2016 Feb 18. PMID 27156759
- [Background] Fenske W, Refardt J, Chifu I, Schnyder I, Winzeler B, Drummond J, Ribeiro-Oliveira A Jr, Drescher T, Bilz S, Vogt DR, Malzahn U, Kroiss M, Christ E, Henzen C, Fischli S, Tonjes A, Mueller B, Schopohl J, Flitsch J, Brabant G, Fassnacht M, Christ-Crain M. A Copeptin-Based Approach in the Diagnosis of Diabetes Insipidus. N Engl J Med. 2018 Aug 2;379(5):428-439. doi: 10.1056/NEJMoa1803760. PMID 30067922
- [Background] Timper K, Fenske W, Kuhn F, Frech N, Arici B, Rutishauser J, Kopp P, Allolio B, Stettler C, Muller B, Katan M, Christ-Crain M. Diagnostic Accuracy of Copeptin in the Differential Diagnosis of the Polyuria-polydipsia Syndrome: A Prospective Multicenter Study. J Clin Endocrinol Metab. 2015 Jun;100(6):2268-74. doi: 10.1210/jc.2014-4507. Epub 2015 Mar 13. PMID 25768671
- [Background] Bolat F, Oflaz MB, Guven AS, Ozdemir G, Alaygut D, Dogan MT, Icagasoglu FD, Cevit O, Gultekin A. What is the safe approach for neonatal hypernatremic dehydration? A retrospective study from a neonatal intensive care unit. Pediatr Emerg Care. 2013 Jul;29(7):808-13. doi: 10.1097/PEC.0b013e3182983bac. PMID 23823259
- [Background] Alshayeb HM, Showkat A, Babar F, Mangold T, Wall BM. Severe hypernatremia correction rate and mortality in hospitalized patients. Am J Med Sci. 2011 May;341(5):356-60. doi: 10.1097/MAJ.0b013e31820a3a90. PMID 21358313
- [Background] Borra SI, Beredo R, Kleinfeld M. Hypernatremia in the aging: causes, manifestations, and outcome. J Natl Med Assoc. 1995 Mar;87(3):220-4. PMID 7731073
- [Background] Darmon M, Pichon M, Schwebel C, Ruckly S, Adrie C, Haouache H, Azoulay E, Bouadma L, Clec'h C, Garrouste-Orgeas M, Souweine B, Goldgran-Toledano D, Khallel H, Argaud L, Dumenil AS, Jamali S, Allaouchiche B, Zeni F, Timsit JF. Influence of early dysnatremia correction on survival of critically ill patients. Shock. 2014 May;41(5):394-9. doi: 10.1097/SHK.0000000000000135. PMID 24667611
- [Background] Andersen LJ, Andersen JL, Pump B, Bie P. Natriuresis induced by mild hypernatremia in humans. Am J Physiol Regul Integr Comp Physiol. 2002 Jun;282(6):R1754-61. doi: 10.1152/ajpregu.00732.2001. PMID 12010758
- [Background] Sands JM, Klein JD. Physiological insights into novel therapies for nephrogenic diabetes insipidus. Am J Physiol Renal Physiol. 2016 Dec 1;311(6):F1149-F1152. doi: 10.1152/ajprenal.00418.2016. Epub 2016 Aug 17. PMID 27534996
- [Background] Gordon CE, Vantzelfde S, Francis JM. Acetazolamide in Lithium-Induced Nephrogenic Diabetes Insipidus. N Engl J Med. 2016 Nov 17;375(20):2008-2009. doi: 10.1056/NEJMc1609483. No abstract available. PMID 27959610
- [Background] Chauhan K, Pattharanitima P, Patel N, Duffy A, Saha A, Chaudhary K, Debnath N, Van Vleck T, Chan L, Nadkarni GN, Coca SG. Rate of Correction of Hypernatremia and Health Outcomes in Critically Ill Patients. Clin J Am Soc Nephrol. 2019 May 7;14(5):656-663. doi: 10.2215/CJN.10640918. Epub 2019 Apr 4. PMID 30948456
- [Background] Muhsin SA, Mount DB. Diagnosis and treatment of hypernatremia. Best Pract Res Clin Endocrinol Metab. 2016 Mar;30(2):189-203. doi: 10.1016/j.beem.2016.02.014. Epub 2016 Mar 4. PMID 27156758
- [Background] Lindner G, Schwarz C, Kneidinger N, Kramer L, Oberbauer R, Druml W. Can we really predict the change in serum sodium levels? An analysis of currently proposed formulae in hypernatraemic patients. Nephrol Dial Transplant. 2008 Nov;23(11):3501-8. doi: 10.1093/ndt/gfn476. Epub 2008 Aug 22. PMID 18723567
- [Background] de Vos EAJ, van der Voort PHJ. ICU acquired hypernatremia treated by enteral free water - A retrospective cohort study. J Crit Care. 2021 Apr;62:72-75. doi: 10.1016/j.jcrc.2020.11.013. Epub 2020 Nov 21. PMID 33285372
- [Background] McCowen KC, Malhotra A, Bistrian BR. Stress-induced hyperglycemia. Crit Care Clin. 2001 Jan;17(1):107-24. doi: 10.1016/s0749-0704(05)70154-8. PMID 11219223
- [Background] Popas RH. Treatment of hypernatremia in adults. In: Emmett M, Forman JP, eds. Wolters Kluwer; 2020. Available at: https://www.uptodate.com
- [Background] Sarahian S, Pouria MM, Ing TS, Sam R. Hypervolemic hypernatremia is the most common type of hypernatremia in the intensive care unit. Int Urol Nephrol. 2015 Nov;47(11):1817-21. doi: 10.1007/s11255-015-1103-0. Epub 2015 Sep 16. PMID 26377488
- [Background] Nur S, Khan Y, Nur S, Boroujerdi H. Hypernatremia: correction rate and hemodialysis. Case Rep Med. 2014;2014:736073. doi: 10.1155/2014/736073. Epub 2014 Nov 9. PMID 25431600
- [Background] Ma F, Bai M, Li Y, Yu Y, Liu Y, Zhou M, Li L, Jing R, Zhao L, He L, Li R, Huang C, Wang H, Sun S. Continuous Venovenous Hemofiltration (CVVH) Versus Conventional Treatment for Acute Severe Hypernatremia in Critically Ill Patients: A Retrospective Study. Shock. 2015 Nov;44(5):445-51. doi: 10.1097/SHK.0000000000000443. PMID 26473438